CLINICAL TRIAL: NCT06581003
Title: Hyperbaric Oxygen Treatment for Veterans With Traumatic Brain Injury
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: James A. Haley Veterans' Hospital (JAHVH) (Unknown)
Responsible Party: Principal Investigator, Harry Van Loveren, Chair Department of Neurosurgery and Brain Repair, University of South Florida
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY006819: HBOT for TBI
Record Dates: First submitted 2024-08-23; First posted 2024-08-30 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-01

CONDITIONS: Traumatic Brain Injury; Military Operations
Keywords: hyperbaric chamber; neuromodulation
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Blinded Group Sequential Adaptive Randomized Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To reduce performance bias participants will blinded to condition. To reduce detection bias, investigators, Independent Evaluators (IE), and data analysts will also be blinded to treatment condition (i.e. HBOT or placebo/sham group). Treatments will be coded in the database (E.g., treatment A or B). Because the primary and secondary outcome data will be collected using a self-report questionnaire, the possibility of interpretation does not exist. Only in case of safety issues, the patient assignment could be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- HBOT Group (Experimental): HBOT chamber pressurized to 2.0 ATA with 100% oxygen
  Interventions: Drug: Oxygen 99.7 %
- Placebo/Sham Group (Sham Comparator): HBOT chamber that remains unpressurized and has 21% oxygen
  Interventions: Drug: Oxygen 21 %

INTERVENTIONS:
Drug: Oxygen 99.7 % — The experimental group will undergo HBOT in a specialized chamber at a pressure of 2.0 ATA. Oxygen will be delivered at 100% for 60 minutes.
  Arms: HBOT Group
Drug: Oxygen 21 % — The control group will be placed in the same specialized chamber, but pressure will be 1.0 ATA (normobaric), and oxygen will be delivered at 21% (normal oxygen concentration in room air) for 60 minutes.
  Arms: Placebo/Sham Group

SUMMARY:
The goal of this blinded, adaptive, randomized, placebo-controlled clinical trial is to investigate the use of hyperbaric oxygen as a therapy to treat mild to moderate traumatic brain injury in Veterans and active military. The main questions it aims to answer are:

* Does Hyperbaric Oxygen Therapy (HBOT) reduce neurobehavioral symptoms? (Aim 1)
* How many HBOT sessions are needed to achieve a significant reduction in neurobehavioral symptoms? (Aim 2)
* Does HBOT reduce posttraumatic stress disorder (PTSD) symptoms? (Aim 3)

Exploratory objectives will explore if there are changes in: 1.) cognitive functioning using neuropsychological tests and the National Institutes of Health (NIH) toolbox, 2.) inflammation biomarkers in blood, 3.) microbiome in stool samples, 4.) electroencephalogram (EEG), 5.) sleep characteristics, and 6.) fMRI.

Research will compare HBOT therapy to a placebo condition to see if HBOT works to treat neurobehavioral symptoms. The placebo condition is a chamber that remains unpressurized and has 21% oxygen.

Participants will:

1. Complete baseline assessments to determine eligibility.
2. Attend 40 sessions of HBOT or placebo (normal air) within 12 weeks.
3. Complete questionnaires and interviews throughout the course of the study.
4. Complete a 2-week post treatment visit

DETAILED DESCRIPTION:
Participants who consent to the study will undergo a comprehensive baseline assessment in two sessions.

Baseline A. This visit will involve questions about the participant's brain injury and relevant medical history, and surveys to learn about symptoms related to the participant's mood, sleep, pain, behaviors (e.g. drug and alcohol use), and life satisfaction. Some surveys may be administered via an interview or as an electronic survey. After Baseline A assessments are completed, the investigators will determine if the participant meets the initial criteria to continue participation.

Baseline B. During this in-person visit, the investigators will have the participant do some thinking exercises by asking him/her to remember words, make decisions about shapes, draw and remember figures, and other similar tasks. The participant will also be asked questions about stress-related symptoms. The investigators will also draw up to 65-mL of blood from the participant's arm to detect inflammation and a brief physical exam (e.g. vision test, breathing functioning, heart rate). The participant will have a chance to complete optional procedure (described below). After Baseline B, the investigators will determine if the participant is eligible to continue their participation. If the participant is eligible, the next stage is "Randomization" to treatment. If the participant is not eligible, study participation will be over.

Randomization: The participant will be randomized to either HBOT (chamber pressurized to 2 ATA with 100% oxygen) or to a placebo condition (chamber that remains unpressurized and has 21% oxygen). The participant will not get to choose the treatment. The participant nor the PI will know which treatment is received.

HBOT or Placebo Dives: Both conditions will take place in a chamber, and each treatment session is called a "dive". The participant will then complete 40 HBOT or placebo dives in 12 weeks at USF. Every dive, the investigators will record the participant's blood pressure, respiration (breathing) rate, and pulse. If the participant is diabetic, the investigators will also record their glucose levels. Then the participant will change into a medical gown and lay down in a clear chamber for their dive. The participant will be in the chamber for about 76 minutes (60 min treatment). Every 5 dives, the participant will complete self-report measures about how they are currently feeling and a barotrauma screening. Every 10 dives, participants will undergo another a brief physical exam, similar to Baseline B. While the FDA has approved HBOT for some conditions, it is considered an experimental therapy for TBI. The entire visit should last about 90 minutes from self-report measures to getting dressed. The participant's regular medical treatment will not change if they take part in the research.

Mid-treatment Assessments: After the 20th dive is complete, the investigators will ask the participant to complete a mid-treatment assessment visit. The investigators do this to monitor how the participant are feeling and thinking. During this visit the participant will complete many of the same self-report measures and interviews as they did during the baseline visits. The participant will also give up to 65-mL of blood at this mid-treatment visit.

Posttreatment Assessments: After the 40 dives are complete, the investigators will ask the participant to complete 1 post-treatment visit at approximately 2 weeks after the last dive. The investigators do this to continue monitoring how the participant is feeling and thinking. During this assessment the participant will complete many of the same self-report measures and interviews as he/she did during the baseline visits and the mid-treatment visit. In addition, the participant will answer a question about global impression of change. They will also be asked to which group they believe they were assigned to: Treatment or Sham. The participant will also give up to 65-mL of blood. After the participant completes the Posttreatments assessments, the investigators will tell him/her which treatment he/she was randomized to receive. If the participant was randomized to the Placebo treatment, he/she will be given the opportunity to receive the actual treatment.

ELIGIBILITY:
Inclusion Criteria:

1. U.S. Service Members and Veterans, between 18 and 75 years of age
2. Ability to read, write, and speak English.
3. Ability to provide informed consent.
4. History of TBI. Participants must have a minimum of 1 year post injury and a TBI classified as mild to moderate as determined by with the Ohio State University TBI Identification Method (Bogner, 2009).
5. Experiencing chronic symptoms of TBI as determined by at least a NSI total score of ≥22 (based on previous work using this score; Harch et al., 2020.
6. Able to tolerate the HBOT environment lying down for one hour.

Exclusion Criteria:

1. Received HBOT within the last 3 months.
2. Concurrently enrolled in another clinical trial.
3. Pregnancy or plans to become pregnant during the study period.
4. Lactating
5. History of retinal repair
6. Malignancy:

   1. Active
   2. Tumor-related chemotherapy within the prior 6 months
   3. Therapeutic radiation to the central nervous system within the prior year
7. Current diagnosis of bipolar disorder type I or schizophrenia as determined by responses to inquiry: Have you ever been diagnosed or prescribed medications for bipolar disorder or schizophrenia?
8. Chronic use of supplemental oxygen or hypoxemia while breathing room air.
9. Untreated asthma/Bronchial obstruction/pulmonary blebs, recent/untreated pneumothorax
10. Congestive heart failure with ejection fraction < 40%
11. Any implanted devices not cleared for hyperbaric pressurization*.
12. Epilepsy and/ or seizures
13. Scuba diving within the previous month
14. Current suicidal intent as measured by ≥ 3 on the Columbia-Suicide Severity Rating Scale Screener
15. Trapped gas observed indicating Bronchospasm present Tension Pneumothorax
16. Evidence of Noncompliant TM (Until corrected)
17. Evidence of Pneumothorax
18. Evidence of Upper Respiratory Tract Infections
19. Signs and symptoms of viral infections, such as high fevers
20. Emphysema with CO2 retention
21. Optic Neuritis
22. Congenital spherocytosis
23. History of middle ear surgery / disorders
24. Pneumocephalus
25. Optional stool samples will not be collected if someone has diarrhea, vomiting, and took antibiotics in the past 30 days.
26. Antabuse because it predisposes to oxygen toxicity.
27. Other medications that would predispose to oxygen toxicity or known to increase drug toxicity will also be excluded. These are: Disulfuram, Acetazolamide, Sulfamylon; bleomycin, cisplatin, and doxyrubicin.
28. Inability to complete MRIs (e.g., claustrophobia, pacemaker, ferromagnetic implants)* Exclusion criteria for fMRI optional sub-study only

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2028-08-15 (Estimated); Study Completion 2029-08-15 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Neurobehavioral Symptoms at 2 weeks Post Intervention | at 2 weeks post treatment
  Measured by the Neurobehavioral Symptom Inventory (NSI). The severity of each symptom on the NSI is measured using a 5-item scale (0-none to 4-very severe) that asks patients to indicate the extent to which each symptom has disturbed them in the previous 2 weeks. The NSI total score is the sum of severity ratings of the 22 symptoms. Cluster scores (domains: physical, cognitive, affective, and sensory) were derived.

SECONDARY OUTCOMES:
Change from Baseline in post traumatic stress disorder symptoms at 2 weeks post intervention | at 2 weeks post treatment
  measured by the PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders - 5 (DSM-5); PTSD Checklist-5 (PCL-5). The PTSD Checklist for DSM-5 (PCL-5) is a self-report measure used to assess the presence and severity of PTSD symptoms based on the criteria in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5). A score between 0-80 Higher Scores: Indicate a worse outcome, as they suggest a greater severity of PTSD symptoms.
  Lower Scores: Indicate a better outcome, as they suggest fewer or less severe PTSD symptom

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ajayi OD, Gaskill Z, Kelly M, Logue CJ, Hendricksen SM. A comparison of two hyperbaric oxygen regimens: 2.0 ATA for 120 minutes to 2.4 ATA for 90 minutes in treating radiation-induced cystitis Are these regimens equivalent? Undersea Hyperb Med. 2020 Fourth Quarter;47(4):581-589. doi: 10.22462/10.12.2020.7. PMID 33227834
- [Background] Daly S, Thorpe M, Rockswold S, Hubbard M, Bergman T, Samadani U, Rockswold G. Hyperbaric Oxygen Therapy in the Treatment of Acute Severe Traumatic Brain Injury: A Systematic Review. J Neurotrauma. 2018 Feb 15;35(4):623-629. doi: 10.1089/neu.2017.5225. Epub 2018 Jan 22. PMID 29132229
- [Background] Loignon A, Ouellet MC, Belleville G. A Systematic Review and Meta-analysis on PTSD Following TBI Among Military/Veteran and Civilian Populations. J Head Trauma Rehabil. 2020 Jan/Feb;35(1):E21-E35. doi: 10.1097/HTR.0000000000000514. PMID 31479073